CLINICAL TRIAL: NCT03377543
Title: Patterns of Sleep Restriction and Recovery: the Inflammatory Resolution Pathways
Brief Title: Sleep and Inflammatory Resolution Pathway
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Monika Haack, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2017P000484
Record Dates: First submitted 2017-12-04; First posted 2017-12-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Response; Inflammation; Sleep; Sleep Restriction
MeSH Terms: conditions — Inflammation | interventions — Aspirin; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control Sleep/Non-Active Placebo or 81mg Aspirin Pill (Experimental): Daily intake of pill at bedtime over 2-week period prior to and during the 11-day in-hospital stay
  Interventions: Drug: Aspirin; Drug: Placebo
- Sleep Restriction/81mg Aspirin Pill (Experimental): Daily intake of pill at bedtime over 2-week period prior to and during the 11-day in-hospital stay
  Interventions: Drug: Aspirin
- Sleep Restriction/Non-Active Placebo (Experimental): Daily intake of pill at bedtime over 2-week period prior to and during the 11-day in-hospital stay
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 81mg aspirin pill daily at bedtime over a 25 day period
  Other Names: Non-steroidal anti-inflammatory drug
  Arms: Control Sleep/Non-Active Placebo or 81mg Aspirin Pill; Sleep Restriction/81mg Aspirin Pill
Drug: Placebo — 81mg non-active pill that looks like aspirin
  Arms: Control Sleep/Non-Active Placebo or 81mg Aspirin Pill; Sleep Restriction/Non-Active Placebo

SUMMARY:
Goal of this project is to investigate whether increases in inflammation that result from common patterns of restricting sleep on week nights and catching up on sleep over the weekend are caused by disruption in the newly discovered inflammatory resolution pathways. These pathways are crucial in the active termination of the inflammatory response, and their disruption may contribute to ongoing unresolved inflammation, which has been observed not only during periods of sleep restriction, but also after recovery sleep has been obtained. If the hypothesis is true, it is possible that increasing the body's natural production of endogenous, inflammatory resolution mediators may provide a non-behavioral strategy to limit the inflammatory consequences in those undergoing periods of sleep restriction with intermittent recovery sleep.

DETAILED DESCRIPTION:
Low-grade or unresolved inflammation is involved in the pathogenesis of many human diseases. Common sleep patterns of restricting sleep during the work week and "catching up" on sleep over the weekend lead to inflammatory upregulation that does not recover completely after the weekend.

The goal of this proposal is to investigate, for the first time, inflammatory resolution pathways. Inflammatory resolution mediators, such as resolvins, are derived from omega-3 free fatty acids and actively 'turn-off' inflammation. Based on preliminary data, the investigators hypothesize that common sleep restriction-recovery patterns disrupt inflammatory resolution pathways, making it difficult to return to inflammatory homeostasis. If true, pharmacologically increasing the body's natural production of endogenous inflammatory resolution mediators may provide a way to reduce the detrimental inflammatory consequences of common sleep restriction-recovery patterns.

The hypothesis will be tested using an experimental model that mimics common patterns of restricting sleep on weekdays and "catching up" on sleep on the weekend. The proposal will further utilize the unique ability of low-dose aspirin, which - like no other non-steroidal anti-inflammatory drug - is able to activate inflammatory resolution pathways. Healthy women and men between the ages of 18 to 65 years will be tested under three, 11-day in-hospital stays, during which participants will be exposed to control sleep or common patterns of sleep restriction-recovery. The three in-hospital stays will be combined with preemptive administration of low-dose aspirin or a placebo.

Targeting inflammatory resolution pathways could provide a novel, non-behavioral strategy to mitigate both inflammatory consequences and future disease risks in those undergoing periods of sleep restriction-recovery patterns - a behavior pattern that is unlikely to be eradicated in the near future, as changes in sleep are generally difficult to make and to maintain.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between the ages 18-65 years.
* Body mass index (BMI) between 18.5 and 35 kg/m2.
* For female participants: No significant discomfort during pre-menses/menses.
* Daily sleep duration between 7-9 hours, verified by electronic sleep diary data for two weeks.
* Habitual sleep period must begin within one hour of 11:00pm (to ensure normal entrainment).
* Negative toxicology screen, including: amphetamines, barbiturates, benzodiazepines, cocaine, opiates, and methadone. Toxicology screening will be performed as part of the screening lab tests; an outside lab toxicology screening will not suffice.

Exclusion Criteria:

* Active infection/disease.
* Following blood chemistry values outside of the laboratory's normal range or the range specified below:

  * WBC (range: 2.0-10.0 K/uL)
  * Platelet count
  * Hematocrit in range
  * TSH outside of the laboratory's normal range
  * Bilirubin >1.5 upper limit of normal
  * ALT or AST >2.5 upper limit of normal
* Stage 4 chronic kidney disease based on CKD epi-equation
* Pre-diabetes or diabetes (HbA1c >5.7%)
* History of neurological, chronic pain, immune/inflammatory, vascular/cardiovascular (including Raynaud syndrome), liver/kidney, metabolic disorders (including diabetes).
* Current asthma (diagnosis of asthma and either asthma symptoms present within the past years or taking medication for asthma) and/or history of ASA induced sensitivity
* Systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90 mmHg prior to the initial and medical screens. Systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg during admissions (Stays 1, 2, and 3)
* History of gastrointestinal disorders, including esophageal reflux, gastric and duodenal ulcers, gastrointestinal bleeding.
* Personal or family (first degree relative) history of any stroke
* History of psychiatric disorders, including major depressive disorders, bipolar disorders, panic disorders, post-traumatic stress disorders (PTSD), thought disorders, and substance abuse/dependence disorders.
* History of intolerance or allergy to non-steroidal anti-inflammatory drugs (NSAID).
* Sleep disorders: Sleep efficiency <80% based on polysomnographic (PSG) screening night; respiratory disturbance index of >10 events/hour based on PSG screening night, periodic leg movement index (PLMI) of >25/hour and/or PLMAI (PLM arousal index) of >5/hour based on PSG screening night; restless legs syndrome, circadian rhythm disorders, and nightmare disorders determined by diagnostic interview.
* Pregnant/nursing.
* Regular medication use other than oral contraceptives.
* Intake of non-steroidal anti-inflammatory drugs (NSAIDs) or cold/cough remedies within the last month.
* Intake of dietary supplements containing DHA/EPA-derived fatty acids (e.g., fish oil) within the last 3 months prior to study start.
* Donation of blood or platelets within three months prior to or in-between study arms.
* Smoking.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Resolution Markers | Change from baseline to sleep restriction, single measure in the morning
  Resolvins

SECONDARY OUTCOMES:
Inflammatory Markers | Change from baseline to sleep restriction, single measure in the morning
  Interleukin-6

CONTACTS AND LOCATIONS:
Overall Officials: Monika Haack, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engert LC, Ledderose C, Biniamin C, Birriel P, Buraks O, Chatterton B, Dang R, Daniel S, Eske A, Reed T, Tang A, Bertisch SM, Mullington JM, Junger WG, Haack M. Effects of low-dose acetylsalicylic acid on the inflammatory response to experimental sleep restriction in healthy humans. Brain Behav Immun. 2024 Oct;121:142-154. doi: 10.1016/j.bbi.2024.07.023. Epub 2024 Jul 21. PMID 39043348